CLINICAL TRIAL: NCT04036500
Title: Sublingual Estradiol Versus Oral Estradiol in Transgender Women
Brief Title: Transgender Estradiol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jenna Sarvaideo, Assistant Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00035015
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Transgender Persons
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Estradiol 1 mg oral first, then Estradiol 1 mg sublingual (Experimental): Subjects will take estradiol 1 mg orally after time 0 blood draw. They will get 7 blood draws at hours 0,1,2,3,4,6,8. A wash-out period of at least one week will allow for complete clearance of the exogenous oral estradiol before testing the pharmacokinetics of sublingual estradiol on the same ten patients in the same manner. On day 2 of study, subject will take estradiol 1 mg sublingually after time 0 blood draw, supervised by a research team member to ensure proper dissolution. Blood will be drawn at hours 0,1,2,3,4,6,8 as on day 1 of study.
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Estradiol — Patients will be given estradiol: 1 mg oral and 1 mg sublingual.

SUMMARY:
Blogs, word-of-mouth, and small studies from the 1990s in the premature ovarian insufficiency and menopause populations have suggested sublingual or transdermal estradiol may be safer and/or more effective than an oral formulation. Sublingual administration entails holding the estrogen tablet under the tongue and allowing it to dissolve, where its absorption is enhanced by the rich vascularization under the tongue. According to Price et al., sublingual administration results in rapid absorption with significantly higher estradiol levels than does comparable oral dosing. This is likely because sublingual administration will bypass metabolism by the intestines and liver. The transdermal route, which also bypasses first-pass metabolism, is not associated with an increased venous thromboembolic risk nor a significant increase in plasma triglycerides or HDL-cholesterol levels. As such, transdermal estrogen is often preferred over oral formulations, although it is relatively expensive and not accessible to many transgender women. Conversely, sublingual administration of estrogen tablets is widely available and could be a cost-effective alternative to transdermal estrogen. However, there are no well-conducted studies that have evaluated the safety and efficacy of sublingual estrogen therapy in the transgender population. This pilot study will elucidate how estrogen levels in the blood change following sublingual versus oral administration of estradiol in transgender women. This data may be used later to design larger studies on safety and efficacy.

Additionally, analyzing a dosage method that patients themselves have tried independently and found effective is also important. This approach incorporates intelligence from the transgender community into our research, creating new knowledge that is supported by data but is founded in existing community insights. Thus, the outcomes of this research have the potential to integrate patient input while also aiding in the development of safety recommendations, with the goal of better caring for our transgender patients.

Primary aim. To establish the pharmacokinetics of sublingual estradiol versus oral estradiol in transgender women.

DETAILED DESCRIPTION:
Patient will plan on being in the Adult Translational Research Unit (A-TRU) for 8 hours. They will be assigned to a suite. They will get 7 blood draws at hours 0,1,2,3,4,6,8 and vitals at the beginning of the visit. Vitals will include height, weight, blood pressure, respiration rate, and pulse. Subject is able to eat while in the A-TRU. Day 1 patient will take estradiol 1 mg ORALLY after time 0 blood draw. The medication will be given by registered nurse. A wash-out period of at least one week will allow for complete clearance of the exogenous oral estradiol before testing the pharmacokinetics of sublingual estradiol on the same ten patients in the same manner. Subject cannot take any hormone replacement therapy between their research appointments. On day 2, subject will take estradiol 1 mg SUBLINGUALLY after time 0 blood draw, supervised by a research team member to ensure proper dissolution. Blood will be drawn at hours 0,1,2,3,4,6,8 as on day 1.

ELIGIBILITY:
Inclusion Criteria:

* Transgender male-to-female
* Naive to hormone therapy
* English speaker
* 18 years of age or older

Exclusion Criteria:

* History of hormone replacement therapy
* Orchiectomy
* Needle phobia
* Serious bleeding condition
* Active deep vein thrombosis, pulmonary embolism or history of these conditions
* Active or recent (e.g., within the past year) arterial thromboembolic disease (e.g., stroke, myocardial infarction)
* Liver dysfunction or disease
* History of breast cancer
* Known sensitivity or allergy to any components of the medications used
* Taking potent CYP3A4 inhibitors or inducers, as determined by team pharmacist
* Taking a medication that may cause additional physical or mental harm if stopped

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender male to female
Enrollment: 11 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenna L Investigator, DO, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 3 months after publication
Access Criteria: IPD will be shared if PI is directly contacted and asked for the above information.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by flyers in clinic waiting room and in clinic physician referrals. Subjects were initially screened over the phone with the screening criteria (n=17). There were 11 eligible subjects. One subject signed a consent form, but was withdrawn prior to initiation of the study.
Pre-assignment Details: After the screening visit in which the pharmacist determined if there was metabolism alternating drugs being taken 10 patients were enrolled.
Period: Overall Study
Arm/Group | Estradiol 1 mg Oral First, Then Estradiol 1 mg Sublingual
Started | 11
Completed | 10
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Estradiol Oral: Subjects will take estradiol 1 mg orally after time 0 blood draw. They will get 7 blood draws at hours 0,1,2,3,4,6,8. A wash-out period of at least one week will allow for complete clearance of the exogenous oral estradiol before testing the pharmacokinetics of sublingual estradiol on the same ten patients in the same manner.
  On day 2 of study, subject will take estradiol 1 mg sublingually after time 0 blood draw, supervised by a research team member to ensure proper dissolution. Blood will be drawn at hours 0,1,2,3,4,6,8 as on day 1 of study.
Arm/Group | Estradiol Oral
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Transgender Woman | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Serum Concentration of Estradiol
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Estradiol 1 mg Oral First, Then Estradiol 1 mg Sublingual: Subjects will take estradiol 1 mg orally after time 0 blood draw. They will get 7 blood draws at hours 0,1,2,3,4,6,8. A wash-out period of at least one week will allow for complete clearance of the exogenous oral estradiol before testing the pharmacokinetics of sublingual estradiol on the same ten patients in the same manner. On day 2 of study, subject will take estradiol 1 mg sublingually after time 0 blood draw, supervised by a research team member to ensure proper dissolution. Blood will be drawn at hours 0,1,2,3,4,6,8 as on day 1 of study.
  Estradiol Tablets: Patients will be given estradiol: 1 mg oral or 1 mg sublingual.
Arm/Group | Estradiol 1 mg Oral First, Then Estradiol 1 mg Sublingual
Number analyzed (Participants) | 10
pg/mL
  Max sublingual serum estradiol | 144 (90)
  Max oral serum estradiol | 35 (8)

2. Primary Outcome: Area Under the Serum Concentration Versus Time Curve
Description: Mean for Area Under the Curve(AUC) for sublingual estradiol.
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Estradiol 1 mg Oral First, Then Estradiol 1 mg Sublingual
Number analyzed (Participants) | 10
mg*h/L | 74.0883 (17.18)

3. Primary Outcome: Oral Clearance of Estradiol
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | Estradiol 1 mg Oral First, Then Estradiol 1 mg Sublingual
Number analyzed (Participants) | 10
mL/hour | NA (NA) — Data analysis could not be successfully completed with variables provided. Lack of variables made proper analysis impossible. Data was below the level of detection.

4. Secondary Outcome: Ratio of Estrone to Estradiol
Description: Descriptive statistics, such as mean for ratio of estrone to estradiol
Time Frame: 8 hours
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Estradiol Oral
Number analyzed (Participants) | 10
Ratio
  estradiol to estrone ratio, sublingual | 1.1 (1)
  estradiol to estrone ratio, oral | 0.7 (0.4)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for an 9 day period (time in which participants were in the study)
Description: 9 days
  1 day of 1mg estradiol orally, 1 week washout, 1 day 1 mg sublingually
Groups:
- Oral Estradiol: Subjects will take estradiol 1 mg orally after time 0 blood draw. They will get 7 blood draws at hours 0,1,2,3,4,6,8. A wash-out period of at least one week will allow for complete clearance of the exogenous oral estradiol.
  Estradiol Tablets: Patients will be given estradiol: 1 mg oral.
- Sublingual Estradiol: On day 2 of study, subject will take estradiol 1 mg sublingually after time 0 blood draw, supervised by a research team member to ensure proper dissolution. Blood will be drawn at hours 0,1,2,3,4,6,8 as on day 1 of study.
  Estradiol Tablets: Patients will be given estradiol: 1 mg sublingually.
Arm/Group | Oral Estradiol | Sublingual Estradiol
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT04036500/Prot_000.pdf
  • Informed Consent Form (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT04036500/ICF_001.pdf